CLINICAL TRIAL: NCT04371224
Title: Randomized Phase II Study of NaliCap (Irinotecan Liposome/Capecitabine) Compared to NAPOLI (Irinotecan Liposome/5-fluorouracil/Leucovorin) in Gemcitabine-pretreated Advanced Pancreatic Cancer
Brief Title: NaliCap (Irinotecan Liposome (Nal-IRI)/Capecitabine) vs. NAPOLI (Nal-IRI/5-FU/LV) ) in Advanced Pancreatic Cancer
Acronym: NaliCap
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Do-Youn Oh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1912-090-1089
Record Dates: First submitted 2020-04-26; First posted 2020-05-01 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Capecitabine; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: randomized phase 2 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NaliCap (Experimental): nal-IRI/Capecitabine
  Interventions: Drug: Irinotecan Liposomal Injection [Onivyde]; Drug: Capecitabine
- NAPOLI (Active Comparator): nal-IRI/5-FU/LV
  Interventions: Drug: Irinotecan Liposomal Injection [Onivyde]; Drug: 5-fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Irinotecan Liposomal Injection [Onivyde] — both arm
  Other Names: nal-IRI
Drug: Capecitabine — NaliCap
  Other Names: xeloda
  Arms: NaliCap
Drug: 5-fluorouracil — NAPOLI
  Other Names: 5FU
  Arms: NAPOLI
Drug: Leucovorin — NAPOLI
  Other Names: LV
  Arms: NAPOLI

SUMMARY:
This is an open label, randomized phase 2 study of NaliCap (irinotecan liposome/Capecitabine) compared to NAPOLI (irinotecan liposome/5-FU/LV) in gemcitabine-pretreated advanced pancreatic cancer patients.

DETAILED DESCRIPTION:
* At the time of initial diagnosis of pancreatic cancer, resectable pancreatic cancer is around 20%, locally-advanced pancreatic cancer is around 25-30%, and the remaining is metastatic pancreatic cancer.
* In metastatic pancreatic cancer, Gemcitabine/Abraxane or FOLFIRINOX 5-fluorouracil/leucovorin/irinotecan/oxaliplatin (FOLFIRINOX) is most commonly used regimen as a palliative 1st-line chemotherapy. In gemcitabine-pretreated pancreatic cancer, irinotecan liposome(nal-IRI)/5-fluorouracil(5FU)/leucovorin(LV)(NAPOLI regimen) improved overall survival of patients compared to 5FU/LV. Now, NAPOLI is standard of care in gemcitabine-pretreated pancreatic cancer.
* Oral 5-FU such as TS-1 is used in gemcitabine pretreated pancreatic cancer patients or 1st-line treatment in gemcitabine-intolerable patients.
* Capecitabine is oral 5-FU, which is commonly used in GI cancers, usually replacing intravenous infusion of 5-FU. It improves patient's convenience not requiring vascular access or hospital admission.
* In NAPOLI regimen, iv 5-FU/LV could be replaced with capecitabine. So far, nal-IRI/Capecitabine combination has not yet been tested.
* Based on these rationale, we plan to conduct the open-label, randomized phase 2 study to assess the safety and efficacy of NaliCap (nal-IRI/Capecitabine) compared to NAPOLI (nal-IRI/5-FU/LV) in patients with gemcitabine-pretreated advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age>20 years at time of study entry
3. Histologically confirmed pancreatic ductal adenocarcinoma
4. Advanced stage (unresectable, recurrent)
5. Gemcitabine-pretreated for advanced pancreatic cancer
6. Eastern Cooperative Oncology Group(ECOG) performance status 0, 1
7. Adequate organ function
8. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects.
9. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product (IP) during the last 3 weeks
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug
4. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
5. Known brain metastasis or spinal cord compression.
6. History of allogenic organ transplantation
7. Cardiac event during past 6 months
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
9. Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive hepatitis B virus (HBV) surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc (hepatitis B core antigen)] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
10. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of IP.
11. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
12. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-free survival was defined as the duration between randomization and disease progression, any cause of death before disease progression, or the last follow-up.The event was defined as disease progression and any cause of death.

SECONDARY OUTCOMES:
Objective response rate | through study completion, an average of 1 year
  Partial response and complete response
Overall survival | From date of randomization until the date of first documented date of death from any cause, whichever came first, assessed up to 12 months
  Overall survival was measured from the randomization to the last follow-up or any cause of death. The event was defined as any cause of death.
Adverse events | through study completion, an average of 1 year
  Common Terminology Criteria for Adverse Events (CTCAE)_ver 5.0 will be used.
QOL: eortc qlq-c30 | through study completion, an average of 1 year
  eortc qlq-c30 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, M.D., PhD., Study Director — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No